CLINICAL TRIAL: NCT00343265
Title: Pilot Randomized Trial of Vaginal Progesterone to Prevent Preterm Birth in Multiple Pregnancy
Brief Title: Vaginal Progesterone Versus Placebo in Multiple Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Calgary Health Region (Other); Juniper Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Sue Ross, Adjunct Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18589; 9427-U0206-47C; 104425
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Multiple pregnancy; Vaginal progesterone; Preterm birth in multiple pregnancy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Progesterone gel
  Interventions: Drug: Vaginal progesterone gel
- 2 (Placebo Comparator): Vaginal gel with no medication
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Vaginal progesterone gel — Vaginal gel once daily
  Arms: 1
Drug: Placebo gel — once daily
  Arms: 2

SUMMARY:
The purpose of this study is to see if daily use of vaginal progesterone will prevent preterm birth in women carrying 2 or more babies.

DETAILED DESCRIPTION:
Women who are pregnant with twins or any higher order multiple will be approached to take part. Women will be randomized to get either vaginal progesterone gel or a placebo gel daily from study entry until 35 6/7 weeks. Women can enter the study between 16 - 20 6/7 weeks. Two hundred women will be recruited to take part. Data will be collected on the women and their infants to see if the active medication prolongs pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed multiple pregnancy
* Ultrasound confirmed minimum of 2 live fetuses
* Gestational age 16-20 6/7 weeks

Exclusion Criteria:

* Placenta previa
* Pre-existing hypertension
* Major fetal anomaly
* Monoamniotic, monozygotic multiples
* Maternal seizure disorder
* History of, or active, thromboembolic disease
* Maternal live disease
* Breast malignancy or pathology
* Progesterone dependent neoplasia
* Plans to move to another city during pregnancy
* Sensitivity to progesterone
* Participation in other clinical trials during the pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Gestational age | Delivery

SECONDARY OUTCOMES:
Proportion of women delivering < 35 weeks | Delivery
Proportion of women delivering < 37 weeks | Delivery
Proportion of women having spontaneous preterm delivery | Delivery
Proportion of women having tocolytic therapy | During pregnancy
Treatment compliance | Delivery
Length of stay for mother and infants | Discharge
Infant morbidity and mortality | Discharge
Birth weight | Birth

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wood, MD, Principal Investigator — University of Calgary; Sue Ross, PhD, Study Director — University of Calgary
Locations (1):
- Calgary Health Region, Calgary, Alberta, Canada

REFERENCES:
- [Result] Wood S, Ross S, Tang S, Miller L, Sauve R, Brant R. Vaginal progesterone to prevent preterm birth in multiple pregnancy: a randomized controlled trial. J Perinat Med. 2012 Nov;40(6):593-9. doi: 10.1515/jpm-2012-0057. PMID 23093256